CLINICAL TRIAL: NCT06481930
Title: A Multicenter Real-world Study of Screening of Cervical Cancer Based on Photoelectric Detection
Status: Not yet recruiting | Type: Observational
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Chief physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: K5505
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Uterine Cervical Cancer; High Grade Squamous Intraepithelial Lesions; Low Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The cervical lesion was detected by fluorescence photoelectricity in the enrolled patients: The enrolled patients were detected with fluorescence photoelectric cervical lesion image detector.
  Interventions: Diagnostic Test: Detection of Cervical Lesions by Fluorescence Photoelectric Image

INTERVENTIONS:
Diagnostic Test: Detection of Cervical Lesions by Fluorescence Photoelectric Image — The enrolled patients underwent fluorescence photoelectric cervical lesion image detection, followed by colposcopy and biopsy to obtain histopathological results. The results of fluorescence photoelectric image detection were compared with histopathological results, and at the same time compared with HPV and TCT results at the time of enrollment.

SUMMARY:
The main purpose of this study is to explore the accuracy and clinical value of fluorescent photoelectric cervical lesion image detector as a screening and shunt tool for cervical lesions through a multi-center, large-sample real-world study with histopathology as the gold standard. The secondary purpose of the study was to verify the coincidence of the fluorescent photoelectric cervical lesion image detector with traditional colposcopic chemical staining.

This study is expected to include 20,000 participants with definite histological results, and compare the specificity and sensitivity, negative predictive value and positive predictive value of three cervical lesion screening methods, such as fluorescent photoelectric cervical lesion image detector, HPV nucleic acid detection and cytology detection. The advantages and disadvantages of fluorescent photoelectric cervical disease image detector, HPV nucleic acid detection and cytology examination were analyzed, and their application scenarios were provided to provide evidence-based medical support for the establishment of comprehensive prevention and treatment system of cervical cancer suitable for China's national conditions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, ≤ 65 years old, with a complete cervix without deformity.
* 2. Have clear cervical cancer screening results, meet HPV16/18 (+) or high-risk HPV (+), and cervical cytology results ≥ ASC-US.
* 3. Fully informed and agreed to participate in the study.
* 4. No history of cervical cancer disease and cancer in other parts.

Exclusion Criteria:

* 1. Cannot meet all Inclusion Criteria.
* 2. There is clear immunosuppression, such as HIV infection or organ transplantation, etc., and the vagina or cervix is in the acute inflammation stage。
* 3. There are serious bleeding diseases or photosensitive diseases such as abnormal coagulation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter, parallel controlled, cross-sectional real-world study based on the population of a hospital gynecology clinic (gynecology clinic/colposcopy room).
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of tissue lesion screening based on photoelectric detection | The data collection time for each subject is approximately 7 days, starting from the day of each subject's enrollment and ending when the pathology report of the cervical tissue biopsy under colposcopy is issued.
  The sensitivity, specificity, positive predictive value and negative predictive value of fluorescence photoelectric cervix lesion image detector were calculated by using CIN 2 + as the gold standard determined by histopathology, and compared with those of HPV and TCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China